CLINICAL TRIAL: NCT00658177
Title: A Randomized, Double-blind, Parallel-group, Placebo-controlled Study Evaluating the Efficacy and Safety of Vardenafil Administered for 12 Weeks in a Flexible-dose Regimen Compared to Placebo in Male Erectile Dysfunction Subjects
Brief Title: Study Evaluating the Efficacy and Safety of Flexible-dose Vardenafil in Subjects With Erectile Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100497
Record Dates: First submitted 2008-04-09; First posted 2008-04-14 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Erectile Dysfunction
Keywords: Erectile dysfunction; Vardenafil
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — 20mg to be taken 1 h prior to sexual intercourse
  Arms: Arm 1
Drug: Placebo — Matching placebo
  Arms: Arm 2

SUMMARY:
Study to investigate the efficacy and safety of Vardenafil

ELIGIBILITY:
Inclusion Criteria:

* Men >/= 18 years of age, with 6 months or longer diagnosis of ED as defined by NIH Consensus statement,
* History of unresponsiveness to sildenafil
* Stable sexual relationship for > 6 month.

Exclusion Criteria:

* Primary hypoactive sexual desire
* History of myocardial infarction, stroke or life-threatening arrhythmia within prior 6 month
* Nitrate therapy
* Other exclusion criteria apply according to the US Product Information

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2003-06; Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Sexual Encounter Profile Question 2 | 12 weeks

SECONDARY OUTCOMES:
Sexual Encounter Profile Question 3 | 12 weeks
Internation Index of Erectile Function-Erectile Function domain | 12 weeks
Safety and tolerability | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer